CLINICAL TRIAL: NCT06169891
Title: A Phase 3, Multicenter, Randomized, Double-blind, Double-dummy, Active-controlled Trial to Evaluate the Efficacy and Safety of Recombinant Anti-IL-1β Humanized Monoclonal Antibody Injection in Chinese Participants With Acute Gout
Brief Title: A Study of Recombinant Anti-IL-1β Humanized Monoclonal Antibody Injection in Chinese Participants With Acute Gout
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSGJ-613-AG-III-01
Record Dates: First submitted 2023-11-30; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Acute Gout
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SSGJ-613 200 mg (Experimental): SSGJ-613 200 mg subcutaneous (s.c) once. The s.c. injection could be administered into the abdomen or thigh. Randomized patients will receive one s.c. injection of SSGJ-613 and placebo matching compound betamethasone injection (0.9% sodium chloride) intramuscularly (i.m.) once, on Day 1. The i.m. injection is recommended to be administered deeply into the gluteal muscle.
  Interventions: Drug: Recombinant Anti-IL-1β Humanized Monoclonal Antibody Injection 200 mg; Other: Placebo
- Compound Betamethasone Injection 1 mL (Active Comparator): Compound betamethasone injection 1 mL intramuscularly (i.m) once. The i.m. injection is recommended to be administered deeply into the gluteal muscle. Randomized patients will receive compound betamethasone injection 1 mL i.m. once and placebo matching SSGJ-613 s.c. once, on Day 1.
  Interventions: Drug: Compound Betamethasone Injection; Other: Placebo

INTERVENTIONS:
Drug: Recombinant Anti-IL-1β Humanized Monoclonal Antibody Injection 200 mg — one s.c. injection of SSGJ-613 once, on Day 1.
  Other Names: SSGJ-613 200 mg
  Arms: SSGJ-613 200 mg
Other: Placebo — Participants will receive Placebo matching Compound Betamethasone Injection to maintain the blinding of the Investigational Medicinal Products.
  Other Names: 0.9% sodium chloride injection
  Arms: SSGJ-613 200 mg
Drug: Compound Betamethasone Injection — 1 mL i.m. once on Day 1
  Arms: Compound Betamethasone Injection 1 mL
Other: Placebo — Participants will receive Placebo matching SSGJ-613 to maintain the blinding of the Investigational Medicinal Products.
  Other Names: PBO
  Arms: Compound Betamethasone Injection 1 mL

SUMMARY:
The purpose of this study is to determine the efficacy and safety of recombinant anti-IL-1β humanized monoclonal antibody injection in Chinese participants with acute gout.

DETAILED DESCRIPTION:
Study SSGJ-613-AG-III-01 is a phase 3, multicenter, randomized, double-blind, double-dummy, active-controlled, parallel-group study examining the effect of recombinant anti-IL-1β humanized monoclonal antibody injection versus compound betamethasone injection in Chinese adult patients with frequent flares of acute gouty arthritis who are contraindicated, intolerant, or lack efficacy to non-steroidal anti-inflammatory drugs (NSAIDs) and/or colchicine. The entire treatment period is 48 weeks, consisting of a double-blind treatment period of 24 weeks and an open treatment period of 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 Years to 75 Years, both male and female.
* BMI ≤35 kg/m2.
* Meeting the American College of Rheumatology (ACR) 2015 criteria for the classification of acute arthritis of primary gout.
* History of ≥ 3 gout flares within the 12 months prior to study randomization.
* Onset of current acute gout flare within 4 days prior to study screening.
* Screening pain intensity of the Target Joint ≥ 50 mm on the 0-100 mm VAS.
* Contraindicated, intolerant or lack efficacy to NSAIDs and/or colchicine.
* Accept uric acid lowering treatment according to the requirements of the protocol.

Exclusion Criteria:

* Gout caused by radiotherapy/chemotherapy, lead, organ transplantation, tumors, etc.
* Evidence/suspicion of infectious/septic arthritis, or other acute inflammatory arthritis.
* Presence of severe renal function impairment.
* Intolerance of subcutaneous and intramuscular injection.
* Known presence or suspicion of active or recurrent bacterial, fungal or viral infection at the time of enrollment.
* History of malignant tumor within 5 years before screening.
* Live vaccinations within 8 weeks prior to the start of the study.
* Use of forbidden therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
The Change in Pain Intensity in the Target Joint From Baseline to 72 Hours Post Dose as Measured on a 0-100 mm Visual Analog Scale (VAS) | 72 hours post-dose
  The change in pain intensity from baseline to 72 hours post dose as measured on a 0-100 mm Visual Analog Scale (VAS): 0= no pain and 100= severe pain. Change from baseline = (post-baseline measurement - baseline).
Time to First New Flare | 12 weeks
  The Kaplan Meier method was used to estimate the median time and 95% CI of the first new flares within 12 weeks after the first administration of each group, as well as the event incidence and 95% CI at 12 weeks.

SECONDARY OUTCOMES:
The Change in Pain Intensity in the Target Joint From Baseline to 6, 24, 48 Hours and 7 Days Post Dose as Measured on a 0-100 mm Visual Analog Scale (VAS) | At 6, 24, 48 hours and 7 Days post-dose
  The change in pain intensity from baseline to 6, 12, 48 hours and 7 days post dose as measured on a 0-100 mm Visual Analog Scale (VAS): 0= no pain and 100= severe pain. Change from baseline = (post-baseline measurement - baseline).
The Time to At Least 50% Reduction of Baseline Pain Intensity in the Target Joint after study drug administration | Up to 48 weeks
  The time to at least 50% reduction in Pain intensity from baseline as measured by Visual Analog Scale (VAS) for each treatment group, is estimated using the Kaplan Meier method. Participants scored their pain intensity in the target joint on a 0-100 mm VAS, ranging from no pain (0) to unbearable pain (100).
The Time to Complete Pain Remission of Baseline Pain Intensity in the Target Joint after study drug administration | Up to 48 weeks
  The time to complete pain remission in Pain intensity from baseline as measured by a 5-point Likert scale for each treatment group, is estimated using the Kaplan Meier method. Participants scored their pain intensity in the target joint on a 5-point Likert scale: None, mild, moderate, severe, extremely severe.
Percentage of Participants with Complete Pain Remission of the Target Joint within 12 weeks after study drug administration | 12 weeks
  Participants scored their pain intensity in the target joint on a 5-point Likert scale: None, mild, moderate, severe, extremely severe.
Time to first use of Rescue Medication | Within 7 days after the first administration, within 7 days after the last acute attack of gout during the double blind treatment period
  The Kaplan Meier method was used to estimate the median time and 95% CI of the first use of Rescue Medication.
Percentage of Participants Taking Rescue Medication After Study Drug Administration and Categories and Dosages of Rescue Medication | 12 weeks, 24 weeks, 48 weeks
Likert scores for target joint pain | 7 days, 12 weeks, 24 weeks
  Patients scored their pain intensity on a 5-point Likert scale (none, mild, moderate, severe, extreme).
Time to First New Flare | 24 weeks, 48 weeks
  The Kaplan Meier method was used to estimate the median time and 95% CI of the first new flares after the first administration of each group, as well as the event incidence and 95% CI.
Percentage of Participants with at least 1 new gout flare | 12 weeks, 24 weeks, 48 weeks
Number of new gout flares | 12 weeks, 24 weeks, 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hejian Zou, MD, Principal Investigator — Shanghai Huanshan Hospital Fudan University-Rheumatology; Qinghong Zhou, MD, Study Director — Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd.

IPD SHARING:
Plan to Share IPD: No